CLINICAL TRIAL: NCT02911324
Title: Cannabinoid Medication for Adults With Obsessive-Compulsive Disorder (OCD)
Brief Title: Cannabinoid Medication for Adults With OCD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Reilly R. Kayser, Resident of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7239
Record Dates: First submitted 2016-09-12; First posted 2016-09-22 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — nabilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nabilone (Experimental): Will receive nabilone at 1 mg daily (BID) over 4 weeks.
  Interventions: Drug: Nabilone
- Nabilone and EX/RP (Experimental): Will receive nabilone at 1 mg daily (BID) plus therapist-guided Exposure and Response Prevention Therapy during 4 weeks.
  Interventions: Drug: Nabilone; Behavioral: Exposure and Response Prevention Therapy

INTERVENTIONS:
Drug: Nabilone — Nabilone is a synthetic cannabinoid that is thought to be a Cannabinoid receptor type 1 (CB 1) agonist. It acts on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD.
  Other Names: Cesamet (brand name)
Behavioral: Exposure and Response Prevention Therapy — Exposure and Response Prevention Therapy (EX/RP) is a type of Cognitive-Behavioral Therapy for OCD that involves intentionally confronting situations that trigger obsessional distress while refraining from doing compulsions.
  Arms: Nabilone and EX/RP

SUMMARY:
The purpose of this pilot research study is to test the effects of a medication called nabilone (Cesamet) in adults with obsessive-compulsive disorder (OCD). Participants will receive either nabilone on its own, or nabilone in combination with a form of cognitive-behavioral therapy (CBT) called exposure and response prevention (EX/RP). Nabilone is a synthetic cannabinoid and acts on the brain's "endocannabinoid system," which has been hypothesized to play a role in OCD. Nabilone is approved by the FDA for the treatment of chemotherapy-induced nausea and vomiting. It is not FDA-approved for treating OCD.

DETAILED DESCRIPTION:
The two first-line treatments for OCD are a class of medications called serotonin reuptake inhibitors (SRIs) and a type of cognitive behavioral therapy called exposure and response prevention (EX/RP). But more than a third of patients with OCD do not respond to these treatments, and less then half become well. Thus, new treatment approaches are needed.

EX/RP is thought to involve fear extinction learning. Recent research suggests that modulators of the endocannabinoid system such as nabilone (a synthetic cannabinoid and agonist of the cannabinoid 1 receptor, CB1R) may enhance fear extinction learning and therefor could enhance EX/RP. However, nabilone could also work via modulating activity in cortico-striatal circuits, which contain high concentrations of CB1R, and thereby might reduce repetitive behaviors like compulsions seen in OCD.

To test both ideas, we will conduct a small pilot randomized trial to explore the effects of nabilone on its own for 4 weeks, vs. combined with EX/RP, in adult patients with OCD. This proof-of-concept study will investigate whether nabilone administration is feasible and well-tolerated in adult patients with OCD. The intent is to collect pilot data to support future grant applications.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Physically healthy, not pregnant
* Primary Obsessive-Compulsive Disorder (OCD)
* Patient off all psychotropic (except selective serotonin reuptake inhibitors [SSRIs]) and other types of drugs likely to interact with nabilone
* Ability to provide informed consent
* Ability to tolerate a treatment free-period

Exclusion Criteria:

* History of any significant medical condition that may increase the risk of participation
* Females who are pregnant or nursing
* Current or lifetime history of psychiatric disorders other than OCD that may increase the risk of participation (e.g. lifetime psychosis or bipolar disorder)
* Current substance use disorder or positive urine toxicology at screening, or any adverse reaction to a cannabinoid
* Patients already receiving EX/RP

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen B Simpson, M.D., Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nabilone | Nabilone and EX/RP
Started | 9 | 7
Completed | 6 | 6
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the nabilone+EX/RP group completed the study, but was not included in the final analysis due to inconsistent self-reporting of symptoms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nabilone | Nabilone and EX/RP | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (14.6) | 30.8 (10.4) | 33.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 3 | 3 | 6
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Yale-Brown Obsessive-Compulsive Scale (YBOCS) [Mean (Standard Deviation); unit: units on a scale] — Measure of OCD symptom severity. Total YBOCS scores are reported. Scores range from 0 - 40, with higher scores representing more severe symptoms.
  units on a scale | 26.5 (4.2) | 25.4 (5.0) | 26.0 (4.3)
Hamilton Depression Rating Scale, 17-Item (HDRS-17) [Mean (Standard Deviation); unit: units on a scale] — Measure of depression symptom severity. Total HDRS-17 scores are reported. Scores range from 0-52, with higher scores representing greater symptom severity.
  units on a scale | 6.5 (5.3) | 5.0 (1.0) | 5.8 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Yale-Brown Obsessive Compulsive Scale
Description: Yale-Brown Obsessive Compulsive Scale (YBOCS) Minimum Value: 0 Maximum Value: 40 Higher scores indicate more severe symptoms
  Change in YBOCS is calculated by subtracting the Week 4 score from the baseline score
Time Frame: Baseline (Week 0) and Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nabilone | Nabilone and EX/RP
Number analyzed (Participants) | 6 | 5
score on a scale
  Week 4 YBOCS Score | 24.0 (6.9) | 14.2 (4.8)
  YBOCS Change | 2.5 (3.6) | 11.2 (3.4)

2. Secondary Outcome: Feasibility of Recruitment
Description: Number of eligible participants recruited per month over a 1 year period.
Time Frame: Through study completion, an average of 1 year.
Population: 16 total participants were recruited for participation in this study
Measure: Number; unit: participants per month
Groups:
- Flow: # of participants enrolled per month
Arm/Group | Flow
Number analyzed (Participants) | 16
participants per month | 0.73

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Nabilone | Nabilone and EX/RP
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 1/9 | 2/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nabilone (N=9) | Nabilone and EX/RP (N=7)
Anxiety (Nervous system disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size and observational design limits generalizability of data

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT02911324/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2016-05-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT02911324/SAP_001.pdf